CLINICAL TRIAL: NCT05407129
Title: Patients and Families Improving Safety in Hospitals by Actively Reporting Experiences (I-SHARE)
Brief Title: Patients and Families Improving Safety in Hospitals by Actively Reporting Experiences
Acronym: I-SHARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Pediatric Research in Inpatient Settings (PRIS) (Unknown)
Responsible Party: Principal Investigator, Alisa Khan, Pediatric Hospitalist/Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-P00042333
Record Dates: First submitted 2022-05-31; First posted 2022-06-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Family Reported Errors and Adverse Events; Health Disparities; Family Safety Reporting; Patient Safety; Voluntary Incident Reporting; Quality Improvement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): This arm is the usual care arm of parents and providers who are randomized to proceed with usual care and are not given the family safety reporting intervention.
- Experimental: Intervention arm (Experimental): This arm is the intervention arm of parents and providers who are randomized to the family safety reporting intervention on the study units.
  Interventions: Behavioral: Family safety reporting intervention

INTERVENTIONS:
Behavioral: Family safety reporting intervention — Family safety reporting intervention for patients/families
  Arms: Experimental: Intervention arm

SUMMARY:
Hospitals ineffectively examine the safety of their processes by relying on voluntary incident reporting (VIR) by clinical staff who are overworked and afraid to report. VIR captures only 1-10% of events, excludes patients and families, and underdetects events in vulnerable groups like patients with language barriers. Patients and families are vigilant partners in care who are adept at identifying errors and AEs. Failing to actively include patients and families in safety reporting and instead relying on flawed VIR presents an important missed opportunity to improve safety. To improve hospital safety, there is a critical need to coproduce (create in partnership with families) effective systems to identify uncaptured errors. Without this information, hospitals are impeded in their ability to improve patient safety. In partnership with diverse families, nurses, physicians, and hospital leaders, investigators created a multicomponent communication intervention to engage families of hospitalized children in safety reporting. The intervention includes 3 elements: (1) a multilingual mobile (email, text, and QR-code) reporting tool prompting families to share concerns and suggestions about safety, (2) family/staff education, and (3) a process for sharing family reports with the unit and hospital so systemic issues can be addressed.

DETAILED DESCRIPTION:
After piloting the intervention in one inpatient unit, marked improvements in family safety reporting and reductions in disparities in reporting by parent education and language results. The investigators now propose to conduct an RCT of the intervention in 4 geographically, ethnically, and linguistically diverse hospitals. The specific aims are to: (1) evaluate the effectiveness of the intervention in improving error detection and other safety outcomes, (2) assess the impact of the intervention on disparities in reporting, and (3) understand contextual factors contributing to successful implementation of the intervention. If effective, the intervention will contribute by: (1) increasing patient/family engagement in reporting, especially from vulnerable groups, (2) identifying otherwise unrecognized events, and (3) enabling hospitals to better understand safety problems in a 360-degree manner and design more effective, patient-centered solutions. Our application has high potential to reshape paradigms for measuring and improving safety and equity.

Hypothesis 1A: The I-SHARE arm will detect higher rates of errors (via I-SHARE tool + VIR) than usual care (via VIR alone).

Hypothesis 1B: In the I-SHARE arm, rates of errors detected by the I-SHARE tool will exceed rates detected through VIR.

Hypothesis 1C: The I-SHARE arm will have higher safety experience, safety climate, and patient activation scores than usual care.

Hypothesis 2A: Among Spanish-speaking and less educated patients/families, the I-SHARE arm will detect higher rates of errors (via I-SHARE tool + VIR) than usual care (via VIR alone).

Hypothesis 2B: In the I-SHARE arm, Spanish-speaking and less educated patients/families will report equal rates of errors as English-speaking and more educated patients/families (via I-SHARE tool).

ELIGIBILITY:
Inclusion Criteria:

* Patient/Family/Caregiver who has been hospitalized on the study unit during the study period (within the past 24 hours) or hospital employee who works at the study sites
* Participants speaking all languages are eligible

Exclusion Criteria:

* Admitted awaiting inpatient psychiatric placement
* In state custody
* Admitted for greater than 24 hours
* Same day discharge
* Covid positive
* Previously enrolled in I-SHARE
* Airborne illness precautions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2028-10-28 (Estimated)

PRIMARY OUTCOMES:
Medical errors | From date of randomization through hospital discharge (typically about 7 days).
  Investigators will evaluate rates and types of errors detected through the mobile tool and through voluntary incident reporting (VIR). Errors will be validated by physician and chart review in real time using an established process the study team has used in prior studies.

SECONDARY OUTCOMES:
Hospital experience | From date of randomization through hospital discharge (typically about 7 days).
  Measured through the Child HCAHPS survey administered prior to discharge. This survey assesses the experience of pediatric patients. It is available in English and Spanish. Particular items of interest include the "preventing mistakes and helping you report concerns" composite measure, which was the single-lowest rated item across hospitals during field testing. This survey consists of closed-ended and Likert scale items. It was developed by the Center of Excellence for Pediatric Quality Measurement at Boston Children's Hospital with funding from AHRQ, CMS, and CHIPRA. The "helping you report" item is assessed on a 3-point scale, with response options of "No," "Yes, somewhat," and "Yes, definitely," with "Yes, definitely" being the best option.
Hospital safety climate | From date of randomization through hospital discharge (typically about 7 days).
  Measured through the Children's Hospital administered prior to hospital discharge Safety Climate Questionnaire (Cox et al. 2013), which contains 14 questions related to parent perceptions of hospital safety climate. Questions were adapted from the AHRQ Hospital Survey on Patient Safety Culture. The survey consists of Likert-scale items and was validated using confirmatory factor analysis. Domains include overall perceptions of safety, staff communication openness, parent communication openness,and handoffs and transitions. This survey is included as a QualityTool in the AHRQ's Health Care Innovations Exchange. Scales range from Strongly Agree to Strongly Disagree (1-5), with Strongly Agree being the best option, except for reverse-coded items, for which Strongly Disagree is the best option.
Patient/parent patient activation | From date of randomization through hospital discharge (typically about 7 days).
  Measured through the PAM (Patient Activation) administered prior to hospital discharge Measure) and the P-PAM (Parent-Patient Activation Measure) to participants. These surveys measure individuals' knowledge, skills, and confidence ("patient activation") in managing their well-being. The 13-item P-PAM was adapted from the PAM measure and is available in English and Spanish and has acceptable validity and reliability in both English and Spanish. The PAM was developed using qualitative methods, Rasch analysis, and test theory psychometric methods. Items on the measure form a unidimensional, probabilistic, Guttman-like scale. Scales range from Strongly Disagree to Strongly Agree (1-4), with Strongly Agree being the best option.
Patient/family reported safety concerns concerns | From date of randomization through hospital discharge (typically about 7 days).
  Will use data from the family safety reporting tool to analyze the percentage of enrolled patient/families that report through the tool. This will allow the team to understand uptake and compare patient/safety reporting among Spanish-speakers vs English-speakers and less educated vs more educated participants enrolled in the intervention arm.

OTHER OUTCOMES:
Patient/family-reported areas for safety improvement | From date of randomization through hospital discharge (typically about 7 days).
  This qualitative outcome is based on a content analysis of patient/family safety reports to identify themes and areas for improvement in real-time that can be shared with the unit and hospital to improve safety.

CONTACTS AND LOCATIONS:
Overall Officials: Alisa Khan, MD, MPH, Principal Investigator — Boston Children's Hospital/Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No